CLINICAL TRIAL: NCT01797497
Title: Parent-Provider Partnerships for Referral Communication
Brief Title: Intervention to Increase Parent-provider Communication During Referrals
Acronym: P3RC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Oklahoma (Other); Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 12-0578; 1 R40MC23632-01-00 (Other Grant/Funding Number: HRSA)
Record Dates: First submitted 2013-02-20; First posted 2013-02-22 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Parent-Provider Communication
Keywords: Parents; Primary Care Providers; Specialists; Children with Special Healthcare Needs; Referral; Health Outcomes; Self-Efficacy; Communication
MeSH Terms: conditions — Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Care plan and coaching group (Experimental): In the intervention group, parents complete a referral care plan with their children's physicians and receive a brief coaching session about how to exchange information with specialists. Outcome data are collected from parents before and after the specialist visit.
  Interventions: Behavioral: Care plan and coaching
- Preintervention group (No Intervention): In the preintervention group, no care plan is used and no coaching takes place. Outcome data are collected from parents before and after the specialist visit.

INTERVENTIONS:
Behavioral: Care plan and coaching — In the intervention group, primary care providers and parents complete their sections of the referral care plan. Parents and referred specialists receive a copy of the form. Parents receive a 5-10 minute brief intervention by phone consisting of education and coaching. The care plan is reviewed with parents to help them practice exchanging information with the specialist and encourage parents to contact their child's primary care provider with any further questions. At the specialist visit, specialists review and complete the care plan with the parent and return the plan to the referring primary care provider. Outcome data are collected from parents before and after the specialist visit.
  Arms: Care plan and coaching group

SUMMARY:
The overall goal of this three-year study is to adapt and test a brief, feasible intervention using a communication tool and brief parent coaching to increase the capability of parents of children and youth with special health care needs to exchange and use medical information in partnership with their child's physicians when their children require sub-specialty referral. We hypothesize that the use of tools to coordinate referrals between physicians and parents will facilitate increased communication between primary care physicians(PCPs) and specialists, and that parents trained in information exchange and care planning will experience increased self-efficacy in interacting with their child's physicians.

There are two primary aims of the study. The first aim is to adapt a joint parent-provider referral communication and care planning intervention (i.e., the 'referral care plan') for use with ethnically diverse populations in an electronic communication environment, and optimize its usability in the practice setting. The second aim is to test the referral care plan in nine pediatric primary care and subspecialty practices in two states, using a stepped wedge cluster randomized trial, to evaluate its effect on communication, parent self-efficacy, and patient outcomes.

DETAILED DESCRIPTION:
One highly-promoted, evidence-based model for chronic illness service delivery for children is the Care Model for Child Health in the Medical Home. The Medical Home (MH) model has been promoted as way to improve quality while making care more efficient. Communication among members of the health care team is an essential part of the model, with sharing of care between providers preferred by families, PCPs and specialists. However, communication between referring and consulting physicians is frequently missing. Failure of communication can produce uncoordinated care, which may contribute to unmet family needs, duplication or omission of needed medical services, and medical errors.

Data on effectiveness of specific MH interventions, especially in children, are scarce. A large intervention in the MH setting was tested using written care plans and use of forms as tools to promote communication with specialists. Results indicated decreases of 40 to 70% in parent reports of lost work/school time, ER visits, and hospital admissions. Additional studies produced decreased hospitalizations and emergency room use in children.

Family-centered care (FCC), a Medical Home core component, has been conceptualized for measurement purposes as having four components: communication with health care providers, shared decision making, providing families with needed information, and self-care management and support. Interventions to improve FCC through parent-to-parent support groups and community-based support have produced increased parent confidence and problem-solving ability. Studies of asthma have shown that teaching primary care providers to take a family-centered approach to medication prescribing as part of an overall education protocol improves symptoms and decreases follow-up visits, and using a family coordinator to help physicians and parents interact more effectively is integral to improving asthma outcomes.

Shared decision-making (SDM), an element of FCC and an approach favored by family advocacy groups to help parents achieve the greatest benefits for their children with special needs, is addressed by our proposed intervention. Merely providing information to patients and families is not sufficient; families must be able to express preferences, participate in dialogue, and make informed decisions as partners with physicians.

The proposed project addresses the health care quality gaps outlined above by improving primary care-specialty-parent communication, family-centered care, and shared decision-making within the MH model. It also addresses knowledge gaps by examining the effectiveness of an important recommended component of the MH and investigating the relationship between the intervention and both process and outcome measures, in a "real-world" practice setting. If the aims of the project are achieved, we will have discovered a practical way to improve care that can be promoted to payers and policymakers.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children aged 0-17, AND
* Parents of children with a chronic health condition, AND
* Parents whose children are receiving a NEW referral to a pediatric neurologist, gastroenterologist, cardiologist, or pulmonologist

Exclusion Criteria:

* Parents of children 18 and older
* Parents of children without a chronic health condition
* Parents of children who are not receiving a referral, or who are receiving a referral to a different sub-specialty

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 97 (Actual)
Dates: Start 2013-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Patient Outcomes | 3 Months
  The main outcome measures of the intervention will be the number of days of lost parent work time or child school time, the number of child ER visits, and the number of unplanned hospital admissions in the 3 months after the specialty visit.

SECONDARY OUTCOMES:
Parent Self-Efficacy | 3 Months
  Self-efficacy in joint treatment planning will be assessed by administering the Perceived Efficacy in Physician-Patient Interactions (PEPPI) scale, a scale originally designed for use to evaluate older persons' self-efficacy in interacting with their physicians that has been successfully used in pediatrics.

OTHER OUTCOMES:
Information Transfer | 3 Months
  Other outcome measures will be accurate information exchange, measured by asking parents and PCPs separately the reason for the child's referral on questionnaires, and asking parents and specialists separately the basic elements of the treatment plan (diagnosis, lab tests planned, and medications if any). A trained specialty nurse clinician reviewer will determine whether parents and physicians agree completely, if they agree partially, or if they disagree. Additionally, for patients in the intervention, parents will be asked whether they have a copy of the care plan (from the PCP) at enrollment and after the specialty visit (completed by the specialist), specialty physicians will be asked whether the care plan was available to them at the time of the consultation, and PCPs will be asked whether the completed care plan was available to them one month after the specialty visit.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Stille, MD, MPH, Principal Investigator — University of Colorado, Denver; Paul Darden, MD, Principal Investigator — University of Oklahoma
Locations (2):
- United States (2):
  - University of Colorado Denver, Denver, Colorado
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma